CLINICAL TRIAL: NCT03005119
Title: A Phase II, Double-blind, Randomized, Placebocontrolled, Parallel-group, Single-center Study to Evaluate the Safety, Tolerability, and Efficacy of Orally Administered PTL201 in Multiple Sclerosis (MS) Patients With Spasticity-related Symptoms
Brief Title: Evaluation of the Safety, Tolerability, and Efficacy of Orally Administered PTL201 in MS Patients With Spasticity-related Symptoms
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PhytoTech Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS-101
Record Dates: First submitted 2016-12-25; First posted 2016-12-29 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTL201 (Experimental): Up to 30 mg/day (30 mg THC, 10 mg CBD), recommended to be administered after meals and if required before bed time. Patients will be instructed not to take more than 10 mg (two capsules) at a single dosing session.
  Interventions: Drug: PTL201
- Placebo (Placebo Comparator): PTL201 and placebo capsules will be identical in appearance
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: PTL201 — Two piece acid resistance hard capsule filled with seamless gelatin matrix green beads containing tetrahydrocannabinol (THC) and cannabidiol (CBD). Each capsule contain 5 mg THC and 5 mg CBD
  Arms: PTL201
Drug: Placebo Oral Capsule — Placebo seamless gelatin matrix green beads containing excipients only
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of oral administration of PTL201 for relief of spasticity-related symptoms in 70 MS patients and to evaluate the efficacy of oral administration of PTL201 in relief of spasticity-related symptoms in MS patients. The pharmacokinetics of PTL201 in comparison to buccally administered Sativex will be evaluated in sub-study prior to the efficacy study.

DETAILED DESCRIPTION:
The study will be comprised of the following parts:

1. Pharmacokinetics (PK) sub-study:

   A 7-day baseline observation period. Randomized cross-over treatments (Sativex, PTL201), performed at minimum 7-day washout.

   Follow up - one week after the last dosing session.
2. Efficacy study:

A 7-day baseline observation period. Single-blind responder phase - 4 weeks. Randomized, double-blind, placebo-controlled treatment phase - 4 weeks Follow up - two weeks.

Subjects participating in the pharmacokinetic sub-study will be allowed to participate in the efficacy study and will not be required to repeat the 7-day observation period of the efficacy study.

Doses will be titrated over a one-week period until reaching maximum tolerated dose (MTD) for each participant The MTD will be self administered for three weeks thereafter. Participants demonstrating response to treatment will continue self administering daily PTL201 treatment or placebo, for an additional four weeks. Participants will keep a daily diary.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (male or female), age 18-65 years
2. Definite diagnosis of MS, according to McDonald 2010 criteria, at least six months prior to enrollment, with MS associated spasticity for at least 3 months prior to enrollment

   1. Patients suffer from moderate to-severe MS-associated spasticity (≥4 sNRS), with no adequate response to traditional antispastic medications
   2. EDSS score: 4 ≤ EDSS ≤ 6; functional motor score ≥3.0 Safety, tolerability and efficacy of PTL201 in reducing multiple sclerosis-associated spasticity-related symptoms
   3. Moderate to severe spasticity in at least two districts of upper and/or lower limbs
3. Anti-spasticity agent(s) and/or disease-modifying medications maintained at a stable dose for 30 days prior to and throughout the study
4. Patients able to self-score spasticity
5. Absence of clinical or neuroradiological relapses from at least three months prior to study entry
6. Willingness and ability to provide written informed consent
7. Willingness and ability to comply with all study requirements
8. Inclusion criteria for placebo-controlled treatment phase:

No major protocol violations were recorded for the patient in the responder phase and at least 20% improvement in sNRS

Exclusion Criteria:

1. Concomitant disease or disorder with spasticity-like symptoms or that may influence the subject's level of spasticity, or medical history suggesting that relapse/remission is likely to recur during the study or expected to influence spasticity
2. Currently using or used cannabis or cannabinoid-based medications within 30 days of study entry and is unwilling to abstain from using them for the duration of the study.
3. Concurrent significant psychiatric, renal, hepatic,cardiovascular or convulsive disorders
4. History or immediate family history of schizophrenia, other psychotic illness, severe personality disorder, or other significant psychiatric disorder other than depression related to MS/MS-associated spasticity.
5. Any known or suspected history of substance abuse/dependence disorder (including opiate abuse),current heavy alcohol consumption, current use of illicit drug, or current non-prescribed use of any prescription drug.
6. Poorly controlled epilepsy or recurrent seizures (i.e., one or more seizures in the past year).
7. Known or suspected hypersensitivity to cannabinoids or to any of the excipients of the study drugs.
8. Myocardial infarction or clinically significant cardiac dysfunction within 12 months of study entry or a cardiac disorder that, in the opinion of the investigator, would put the patient at risk of a clinically significant arrhythmia or myocardial infarction
9. Female patients of child-bearing potential and male patients whose partner is of childbearing potential, unless willing to ensure that they or their partner use effective contraception throughout the study and for three months thereafter
10. Female patient who is pregnant, lactating, or planning pregnancy during the course of the study or within the 3 months thereafter.
11. Any other significant diseases or disorder, which, in the opinion of the investigator, participation in the study may either put the patient at risk or may influence the result of the study, or the patient's ability to participate in the study.
12. Travel outside the country planned during the study.
13. Unwilling to abstain from donating blood during the study.
14. Patients previously randomized into a cannabinoid-based clinical trial for MS pain and spasticity within 6 months of study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of study treatment-related adverse events (AE) | 10 weeks (70 days) from beginning of treatment to end of follow-up
Change in sNRS scores from randomization to end of placebo-controlled treatment phase | during the 4 weeks (28 days) placebo-controlled treatment period

SECONDARY OUTCOMES:
Incidence of all AEs | during 10 week treatment plus follow up period
Percent change in walking velocity | during 4 weeks placebo-controlled treatment period
Clinical Global Impression Improvement (CGI-I) assessment using a 7-point scale condition | at randomization (day 29) and the end of placebo-controlled treatment phase (day 57)
Cadence (steps/min) assessment | at baseline (day 1) end of responder phase (day 29) and end of placebo-controlled treatment phase (day 57)
Stride length (cm) assessment | at baseline (day 1) end of responder phase (day 29) and end of placebo-controlled treatment phase (day 57)
pNRS assessment | at baseline (day 1) end of responder phase (day 29) and end of placebo-controlled treatment phase (day 57)
Spasm frequency assessment | at baseline (day 1) end of responder phase (day 29) and end of placebo-controlled treatment phase (day 57)
Sleep disturbance assessment | at baseline (day 1) end of responder phase (day 29) and end of placebo-controlled treatment phase (day 57)
Assessment of clinical gait measures | at baseline (day 1) end of responder phase (day 29) and end of placebo-controlled treatment phase (day 57)
  Timed (sec) 25 foot walk test (T25FW)
Assessment of clinical gait measures | at baseline (day 1) end of responder phase (day 29) and end of placebo-controlled treatment phase (day 57)
  Timed (sec) up and go test (TUG)

OTHER OUTCOMES:
Combined modified Ashworth score (cMAS) and MS walking scale 12 (MSWS-12) assessments, posturography measure, Selected spatio-temporal parameters of gait | at baseline (day 1) end of responder phase (day 29) and end of placebo-controlled treatment phase (day 57)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba medical center, Tel Hashomer, Ramat Gan, Israel